CLINICAL TRIAL: NCT06635070
Title: The Relationship Between Education Status and Care Burden of Mothers of Individuals With Cerebral Palsy
Status: Not yet recruiting | Type: Observational
Sponsor: Muş Alparslan University (Other)
Responsible Party: Sponsor
Other Study IDs: Cerebral Palsy
Record Dates: First submitted 2024-10-07; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Caregiver Burden; Mother; Educational Status
MeSH Terms: conditions — Cerebral Palsy; Caregiver Burden

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study, examines how maternal education affects caregiving burdens for children with cerebral palsy. Cerebral palsy requires long-term, intensive care, often leading to significant physical, emotional, and financial strain on caregivers. The study aims to assess whether higher maternal education is associated with lower care burdens, possibly due to increased access to resources or coping strategies, and whether lower educational levels result in greater challenges. A survey, combined with standardized measures such as the Caregiver Burden Scale, will be used to quantify the caregiving burden. The results are expected to inform policies or interventions aimed at reducing caregiver strain.

DETAILED DESCRIPTION:
This study titled "The Relationship Between the Education Status of Mothers and the Care Burden of Individuals with Cerebral Palsy" aims to explore how the education level of mothers influences their caregiving responsibilities and burdens while caring for individuals with cerebral palsy. Cerebral palsy, a neurological disorder affecting movement and muscle tone, often requires lifelong caregiving, which can be physically, emotionally, and financially demanding.

The study seeks to investigate whether mothers with higher levels of education experience lower care burdens due to greater access to resources, knowledge of coping strategies, or better healthcare utilization. Conversely, the study will also examine if mothers with lower educational attainment face more significant challenges due to limited access to support systems or information.

The research will involve a mixed-methods approach, including a survey to assess the education level of mothers and the care burden they experience. Specific tools to measure care burden, such as the Caregiver Burden Scale, will be employed. The findings aim to provide insights into the role of education in mitigating caregiving challenges and inform potential interventions or policies that could support caregivers in these situations.

ELIGIBILITY:
Inclusion Criteria:

* Having a child who is receiving education in special education institutions
* The child's diagnosis was made at least 6 months ago
* The disabled individuals must be between the ages of 0-18

Exclusion Criteria:

-

Ages: 20 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Mothers of individuals with cerebral palsy
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-10-21 (Estimated); Primary Completion 2024-12-09 (Estimated); Study Completion 2024-12-16 (Estimated)

PRIMARY OUTCOMES:
Zarit Caregiver Burden Interview | one month
  This scale was developed to assess the stress experienced by those who provide care to a person in need of care or to an elderly person. This scale can be completed by the caregivers themselves or by the researcher. It consists of 22 questions that determine the effect of caregiving on the person's life. The items in the scale are mostly emotional and social. The Turkish validity and reliability were made by Özer et al. in 2006. The scale is graded on a score of 0-4 for each question. Verbal use in the survey is never, rarely, sometimes, often, almost always. Total scores between 0-21 are classified as low or none, between 21-40 as mild or moderate, between 41-60 as moderately severe, and between 61-88 as severe burden. A high scale score indicates that the caregiver is experiencing a lot of distress.